CLINICAL TRIAL: NCT03805373
Title: Validation of a Diet Risk Screening Tool
Acronym: DRS
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: PKE DRS; 19PRE34450165 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2018-12-19; First posted 2019-01-15 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Nutrition; Diet Modification; Preventive Medicine; Cardiovascular Diseases; Health Promotion
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diet Assessment Survey — Participants will complete 2 different diet assessment tools separated by at least 1 week.

SUMMARY:
Cardiovascular disease (CVD) is responsible for 1 in 4 deaths in the US annually. Nutrition is an important part of prevention and management of CVD and other chronic diseases, but only about 25% of patients with a chronic disease diagnosis (and about 12% of patients without a chronic disease) receive nutrition counseling from their physician. The investigators plan to validate a diet questionnaire in preparation for the creation of a diet assessment/ intervention tool to increase rates of nutrition intervention in medical care. The aim of this project is to test whether the developed questionnaire accurately identifies individuals at high nutritional risk compared to the Healthy Eating Index- 2015 (HEI-2015) determined by a validated questionnaire.

DETAILED DESCRIPTION:
Heart disease is the leading cause of death in the US. The risk of heart disease increases with diabetes, overweight/obesity and unhealthy lifestyle behaviors. Despite the well recognized benefits of a healthy lifestyle in reducing heart disease risk, nutrition is not a part of routine medical care. Only about 25% of patients with a chronic disease, such as CVD (and only about 12% of those without a chronic disease), receive nutrition education from their doctor. Doctors often report a lack of confidence in providing nutrition education, and a lack of time in the office visit. Doctors need resources to assess diet and discuss nutrition with patients. This research aims to provide doctors with a diet assessment/ intervention tool to improve rates of nutrition intervention in medical care.

There are few nutrition assessment tools appropriate for use in a medical office visit. The investigators have created a 9-item questionnaire that doctors can use to quickly assess diet in the office visit and plan test to it ensure that it measures diet accurately. In this study, the investigators will test the new questionnaire against an established, validated tool called a food frequency questionnaire. The investigators will also create talking points that physicians can use to help their patients make healthy dietary changes. In the future, the investigators will create a cell phone app based on the questionnaire that can be accessed quickly in an office visit. The app will provide a risk score and personalized talking points that can be discussed with the patient or e-mailed to them directly.

An increase of just 1 serving of fruit per day (1 small apple, 1 cup of berries, 1 orange) could save over 1 million lives per year and reduce heart disease risk dramatically. This project could help to improve nutrition counseling by physicians during office visits, and can be expected to reduce heart disease rates and increase quality of life for those living with heart disease. This is important not only because of the statistics above, but also because when physicians do discuss healthy lifestyle changes with their patients, patients are more likely to make changes and improve their cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* Adults across the United States, ages 35-75, with a computer and Internet access

Exclusion Criteria:

* Any individuals not meeting the study inclusion criteria or not willing to adhere to the study protocol

Ages: 35 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults across the United States, ages 35-75, with a computer and Internet access.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Healthy Eating Index (HEI-2015) Score | Usual intake over the course of 1 week.
  Assess the agreement between DRS (scored out of 27) and HEI-2015 (scored out of 100 points) calculated from Viocare Food Frequency Questionnaire (FFQ)

SECONDARY OUTCOMES:
Servings of prepared foods | Usual intake over the course of 1 week.
  Individual items on the test questionnaire will be validated through comparison to detailed diet data captured in the VioScreen instrument to determine where the questionnaire can be improved (DRS prepared foods=0-3 points, FFQ =0-10 points).
Servings of breads, rolls, sandwiches | Usual intake over the course of 1 week.
  Individual items on the test questionnaire will be validated through comparison to detailed diet data captured in the VioScreen instrument to determine where the questionnaire can be improved (DRS breads/rolls/sandwiches=0-3 points, FFQ=0-10 points).
Servings of salty snacks | Usual intake over the course of 1 week.
  Individual items on the test questionnaire will be validated through comparison to detailed. diet data captured in the VioScreen instrument to determine where the questionnaire can be improved (DRS salty snacks=0-3 points, FFQ=0-10 points).
Servings of processed meats | Usual intake over the course of 1 week.
  Individual items on the test questionnaire will be validated through comparison to detailed. diet data captured in the VioScreen instrument to determine where the questionnaire can be improved (DRS processed meats=0-3 points, FFQ =0-10 points).
Servings of sugar-sweetened beverages | Usual intake over the course of 1 week.
  Individual items on the test questionnaire will be validated through comparison to detailed. diet data captured in the VioScreen instrument to determine where the questionnaire can be improved (DRS sugar-sweetened beverages=0-3 points, FFQ=0-10 points).
Servings of nuts, seeds, nut butters | Usual intake over the course of 1 week.
  Individual items on the test questionnaire will be validated through comparison to detailed. diet data captured in the VioScreen instrument to determine where the questionnaire can be improved (DRS nuts/seeds/nut butters=0-3 points, FFQ=0-10 points).
Servings of fish or shellfish | Usual intake over the course of 1 week.
  Individual items on the test questionnaire will be validated through comparison to detailed. diet data captured in the VioScreen instrument to determine where the questionnaire can be improved (DRS fish/shellfish=0-3 points, FFQ=0-10 points).
Servings of non-starchy vegetables | Usual intake over the course of 1 week.
  Individual items on the test questionnaire will be validated through comparison to detailed. diet data captured in the VioScreen instrument to determine where the questionnaire can be improved (DRS non-starchy vegetables=0-3 points, FFQ=0-10 points).
Servings of fruit | Usual intake over the course of 1 week.
  Individual items on the test questionnaire will be validated through comparison to detailed. diet data captured in the VioScreen instrument to determine where the questionnaire can be improved (DRS fruit=0-3 points, FFQ=0-10 points).

CONTACTS AND LOCATIONS:
Overall Officials: Penny Kris-Etherton, PhD, Principal Investigator — Penn State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Micha R, Penalvo JL, Cudhea F, Imamura F, Rehm CD, Mozaffarian D. Association Between Dietary Factors and Mortality From Heart Disease, Stroke, and Type 2 Diabetes in the United States. JAMA. 2017 Mar 7;317(9):912-924. doi: 10.1001/jama.2017.0947. PMID 28267855
- [Result] Greenwood JL, Lin J, Arguello D, Ball T, Shaw JM. Healthy eating vital sign: a new assessment tool for eating behaviors. ISRN Obes. 2012 Jul 22;2012:734682. doi: 10.5402/2012/734682. eCollection 2012. PMID 24533209
- [Result] Kris-Etherton PM, Akabas SR, Bales CW, Bistrian B, Braun L, Edwards MS, Laur C, Lenders CM, Levy MD, Palmer CA, Pratt CA, Ray S, Rock CL, Saltzman E, Seidner DL, Van Horn L. The need to advance nutrition education in the training of health care professionals and recommended research to evaluate implementation and effectiveness. Am J Clin Nutr. 2014 May;99(5 Suppl):1153S-66S. doi: 10.3945/ajcn.113.073502. Epub 2014 Apr 9. PMID 24717343
- [Derived] Johnston EA, Petersen KS, Beasley JM, Krussig T, Mitchell DC, Van Horn LV, Weiss R, Kris-Etherton PM. Relative validity and reliability of a diet risk score (DRS) for clinical practice. BMJ Nutr Prev Health. 2020 Oct 8;3(2):263-269. doi: 10.1136/bmjnph-2020-000134. eCollection 2020 Dec. PMID 33521537